CLINICAL TRIAL: NCT06670417
Title: Low-level Laser Therapy Versus Offloading Exercises on Foot Ulcer Healing in Patients with Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba afifi, lecturer Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004287
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: Low level laser; Diabetic Foot Ulcer; Blood glucose level
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (A) (Experimental A): will receive extravascular low level laser therapy LLLT (laser watch dev (Experimental)
  Interventions: Device: Low level laser therapy watch: The laser watch device was a semiconductor LLL therapeutic apparatus, (model:SL-03 GaALAs semiconductor) Domer Laser Therapy Watch class 3B 650nm low-level laser light
- B) (Experimental B): will receive Offloading exercise inform of burger allen exercise combined with (Experimental)
  Interventions: Other: Buerger Allen exercise
- (C) Control group will receive their prescribed hypoglycaemic medications(oral and insulin) and usua (Experimental)
  Interventions: Other: Regular wound care

INTERVENTIONS:
Device: Low level laser therapy watch: The laser watch device was a semiconductor LLL therapeutic apparatus, (model:SL-03 GaALAs semiconductor) Domer Laser Therapy Watch class 3B 650nm low-level laser light — Low level laser therapy watch:
  The laser watch device was a semiconductor LLL therapeutic apparatus, (model:SL-03 GaALAs semiconductor) Domer Laser Therapy Watch class 3B 650nm low-level laser light. It provides 18 individual laser beams used for extravascular blood irradiation (transcutaneous) through radial and ulnar vessels at the wrist site.
  Arms: Group (A) (Experimental A): will receive extravascular low level laser therapy LLLT (laser watch dev
Other: Buerger Allen exercise — Procedure-Keep the Buerger Allen exercise board on the cot. Elevate the lower extremities to an angle of 45 to 90 degree with the help of exercise board. Provided support to the lower extremities to maintain the position. Make the subject to maintain the same position in the same manner until the skin blanches (appears dead white). Lower the feet and the legs below the level of the rest of the body until redness appears (care should be taken that there is no pressure against the back of the knees). Place the legs flat on the bed for a few minutes. Ask the subjects to sit in a relaxed position while each foot is flexed and extended then inverted and everted for 3 minutes till the feet turns entirely pink. Ask the subject to rotate the feet in all the direction. Make the subject to lie quietly for 5 minutes, keeping legs warm with a blanket
  Arms: B) (Experimental B): will receive Offloading exercise inform of burger allen exercise combined with
Other: Regular wound care — Regular wound care and dressing to the wound and ulcer
  Arms: (C) Control group will receive their prescribed hypoglycaemic medications(oral and insulin) and usua

SUMMARY:
The goal of this clinical trial is to evaluate the effect of extravascular Low-level laser therapy (LLLT) versus offloading exercises on foot ulcers healing (DFUs) in type 2 diabetic patients. could include sixty patients with type 2 diabetes associated with diabetic foot ulcer as a complication, their ages ranging from 45 - 55 years. Patients will be selected from Faculty of Medicine (Kasr Al-Aini) Cairo University. They will be referred by the physician after a complete medical evaluation. . The main question it aims to answer is there any significant difference between extravascular low-level laser therapy and offloading exercise on diabetic foot ulcer healing in type 2 diabetic patients ?

After clinical assessment patients will be randomly allocated into three groups equal in number:

Group (A) (Experimental A): will receive extravascular low level laser therapy LLLT (laser watch device) combined with their prescribed hypoglycaemic medications(oral and insulin) and usual wound care for 12 weeks (3 sessions/ week).

Group (B) (Experimental B): will receive Offloading exercise inform of burger allen exercise combined with their prescribed hypoglycaemic medications(oral and insulin) and usual wound care for 12 weeks (3 sessions/ week).

Group (C) Control group will receive their prescribed hypoglycaemic medications(oral and insulin) and usual wound care only for 12 weeks (3 sessions/ week).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 25-34.9 kg/m2.
* Glycated hemoglobin (HbA1c) >7 %.
* ABP index absolute normal (1-1.3)
* Patient with polyneuropathy.
* Patient suffer from diabetes more than 5 years.
* Patient has chronic unhealed diabetic ulcer from 4 weeks up to 6 weeks.

Exclusion Criteria:

* Patients with history of hypo- hyperglycemic coma.
* Uncontrolled cardiovascular complications.
* Malignancy, Anemia, Hemorrhagic diseases.
* Cardiac peace maker.
* Deep venous thrombosis.
* Osteomyelitis.
* Patients with Monckeberg sclerosis.
* Photosensitivity to laser.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
wound surface area | From enrollment to the end of treatment at 2 weeks
Glycated hemoglobin HbA1c | From enrollment to the end of treatment at 12weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No